CLINICAL TRIAL: NCT03566823
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Study of SHP647 as Induction Therapy in Subjects With Moderate to Severe Crohn's Disease (CARMEN CD 306)
Brief Title: Efficacy and Safety Study of Ontamalimab as Induction Therapy in Participants With Moderate to Severe Crohn's Disease (CARMEN CD 306)
Acronym: CARMEN CD 306
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to discontinue the SHP647 (ontamalimab) clinical trial development program for inflammatory bowel diseases (IBD) early.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP647-306
Record Dates: First submitted 2018-05-09; First posted 2018-06-25 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — ontamalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ontamalimab 25 mg (Experimental): Participants will receive 25 mg of ontamalimab subcutaneous injection using a prefilled syringe on Week 0/Day 1, Week 4, Week 8, and Week 12.
  Interventions: Biological: Ontamalimab
- Ontamalimab 75 mg (Experimental): Participants will receive 75 mg of ontamalimab subcutaneous injection using a prefilled syringe on Week 0/Day 1, Week 4, Week 8, and Week 12.
  Interventions: Biological: Ontamalimab
- Placebo (Placebo Comparator): Participants will receive placebo matching with ontamalimab subcutaneous injection using a prefilled syringe on Week 0/Day 1, Week 4, Week 8, and Week 12.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ontamalimab — Subcutaneous injection of ontamalimab will be administered using a prefilled syringe.
  Other Names: SHP647; PF-00547659
  Arms: Ontamalimab 25 mg; Ontamalimab 75 mg
Other: Placebo — Subcutaneous injection of placebo matched with ontamalimab will be administered using a prefilled syringe.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ontamalimab in inducing clinical remission and endoscopic response in participants with moderate to severe Crohn's Disease.

DETAILED DESCRIPTION:
27Mar2020: Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic .

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between greater than or equal to (> =) 16 and less than or equal to (<=) 80 years of age; participants less than (<) 18 years of age must weigh >=40 kg and must have body mass index >=16.5 kilogram per meter square (kg/m^2)
* Participants must have active moderate to severe ileal (terminal ileum), ileocolic, or colonic CD at baseline (Visit 2) as defined by:

  1. CDAI score between 220 and 450 (inclusive) AND
  2. Meeting the following subscores in the 2 item PRO:

  i. Abdominal pain subscore >= 5 (average worst daily pain on the 11 point NRS) and abdominal pain subscore >= 2 (average daily pain on the 4-point abdominal pain variable of CDAI) over the 7 most recent days out of the 10 days before colonoscopy preparation (may or may not be contiguous) AND/OR ii. Average of the daily stool frequency subscore >=4 of type 6/7 (very soft stools/liquid stools) as shown in the BSFS over the 7 most recent days out of the 10 days before colonoscopy preparation (may or may not be contiguous) c. Presence of ulcerations that are characteristic to CD, as determined by a colonoscopy performed during screening, and as defined by the SES-CD >6 (SES CD >=4 for isolated ileitis) Note that the participant must be confirmed as meeting the CDAI score and PRO subscore requirements before a colonoscopy is done
* Participants must have a documented diagnosis (endoscopic with histology) of CD for >=3 months before screening. Documented diagnosis is defined as:

  1. A biopsy report in which the description of the histological findings is consistent with the CD diagnosis AND
  2. A report documenting disease duration based upon prior colonoscopy Note: If a biopsy report is not available in the source document at the time of screening, a biopsy must be performed during the screening colonoscopy and the histology report should be consistent with the CD diagnosis. If the histology description does not support the CD diagnosis at this time point, the participant should not be randomized
* Participants must be willing and able to undergo a colonoscopy during screening after all other inclusion criteria have been met
* Participants must have had an inadequate response to, or lost response to, or had an intolerance to at least 1 conventional treatment such as sulfasalazine or mesalamine (5-aminosalicylic acid [5-ASA]), glucocorticoids, or immunosuppressants (azathioprine [AZA], 6-mercaptopurine [6-MP] or methotrexate [MTX]) or anti-tumor necrosis factor (anti-TNF). Participants who have had an inadequate response to sulfasalazine or mesalamine should have also failed at least 1 other conventional treatment such as glucocorticoids
* Participants receiving any treatment(s) for CD are eligible provided they have been, and are anticipated to be, on a stable dose for the designated period of time
* Participants are males or nonpregnant, nonlactating females who, if sexually active, agree to comply with the contraceptive requirements of the protocol, or females of nonchildbearing potential. Males and females of reproductive potential who are sexually active must agree to use appropriate contraception (ie, highly effective methods for female and medically appropriate methods for male study participants, for the duration of the study

Exclusion criteria:

* Participants with indeterminate colitis, microscopic colitis, nonsteroidal anti-inflammatory drug-induced colitis, ischemic colitis, infectious colitis, or clinical/histologic findings suggestive of UC
* Participants with colonic dysplasia or neoplasia. (Participants with prior history of adenomatous polyps will be eligible if the polyps have been completely removed)
* Participants with past medical history or presence of toxic megacolon
* Participants with presence of enterovesical (ie, between the bowel and urinary bladder) or enterovaginal fistulae
* Participants with current symptomatic diverticulitis or diverticulosis
* Participants with clinically significant obstructive colonic stricture, or who have a history of bowel surgery within 6 months before screening, or who are likely to require surgery for CD during the treatment period. Participants who have undergone previous colonic resection or ileocolectomy more than 6 months before screening must have at least 25 cm of colon remaining
* Participants with past medical history of multiple small bowel resections resulting in clinically significant short bowel syndrome
* Participants requiring total parenteral nutrition
* Participants with past medical history of bowel surgery resulting in an existing or current stoma. Participants who had a j-pouch are excluded as a j-pouch could result in a stoma
* Participants have had prior treatment with ontamalimab (formerly PF-00547659; SHP647)
* Participants with known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients
* Participants have received any nonbiologic treatment with immunomodulatory properties (other than AZA, 6-MP, or MTX) or continuous antibiotics (>2 weeks) for the treatment of CD within 30 days before baseline (Visit 2)
* Participants have received anti-TNF treatment within 60 days before baseline (Visit 2)
* Participants have received any biologic with immunomodulatory properties (other than anti-TNFs) within 90 days before baseline (Visit 2)
* Participants have ever received anti-integrin/adhesion molecule treatment (eg, natalizumab,vedolizumab, efalizumab, etrolizumab, or any other investigational anti-integrin/adhesion molecule)
* Participants have received lymphocytes apheresis or selective monocyte granulocytes apheresis within 60 days before baseline (Visit 2)
* Participants have received enteral nutrition treatment within 30 days before baseline (Visit 2)
* Participants have received parenteral or rectal glucocorticoids or rectal 5-ASA within 14 days before screening colonoscopy
* Participants have taken >20 milligram per day(mg/day) of prednisone, >9 mg/day of budesonide, or equivalent oral systemic corticosteroid dose within 14 days before baseline (Visit 2) or have taken >=40 mg/day of prednisone or equivalent oral systemic corticosteroid dose within 6 weeks before baseline (Visit 2)
* Participants have participated in other investigational studies within either 30 days or 5 half-lives of investigational product used in the study (whichever is longer) before screening (Visit 1)
* Participants have received a live (attenuated) vaccine within 30 days before the baseline visit (Visit 2)
* Participants with active enteric infections (positive stool culture and sensitivity), Clostridium difficile infection or pseudomembranous colitis (subjects with C. difficile infection at screening may be allowed retest after treatment), evidence of active cytomegalovirus infection or Listeria monocytogenes, known active invasive fungal infections such as histoplasmosis or parasitic infections, clinically significant underlying disease that could predispose the subjects to infections, or a history of serious infection (requiring parenteral antibiotic and/or hospitalization) within 4 weeks before the baseline visit (Visit 2)
* Participants with abnormal chest x-ray or other imaging findings at screening (Visit 1), such as presence of active tuberculosis (TB), general infections, heart failure, or malignancy (A chest x-ray, computed tomography scan, etc, performed up to 12 weeks before study entry [screening, Visit 1] may be used if available; documentation of the official reading must be located and available in the source documentation)
* Participants with evidence of active or latent infection with Mycobacterium tuberculosis (TB) or participants with this history who have not completed a generally accepted full course of treatment before baseline (Visit 2) are excluded all other participants must have either the Mantoux (purified protein derivative [PPD]) tuberculin skin test or interferon-gamma release assay (IGRA) performed

Participants who have no history of previously diagnosed active or latent TB are excluded if they have a positive Mantoux (PPD) tuberculin skin test (ie >= 5 millimeter [mm] induration) or a positive IGRA (the latter to be tested at the site's local laboratory) during screening or within 12 weeks before screening If the IGRA cannot be performed locally, a central laboratory may be used, with prior agreement from the sponsor:

1. An IGRA is strongly recommended for participants with a prior Bacillus Calmette-Guérin vaccination but may be used for any participant Documentation of IGRA product used and the test result must be in the participant's source documentation if performed locally Acceptable IGRA products include QuantiFERON-TB Gold Plus In-Tube Test
2. If the results of the IGRA are indeterminate, the test may be repeated, and if a negative result is obtained, enrollment may proceed In participants with no history of treated active or latent TB, a positive test on repeat will exclude the participantParticipants with a history of active or latent TB infection must follow instructions for "Participants with a prior diagnosis of active or latent TB are excluded unless both of the following criteria are met" in this criterion
3. Participants with repeat indeterminate IGRA results, with no prior TB history, may be enrolled after consultation with a pulmonary or infectious disease specialist who determines low risk of infection (ie, participant would be acceptable for immunosuppressant [eg, anti-TNF] treatment without additional action) This consultation must be included in source documentation Results from a chest x-ray, taken within the 12 weeks before or during screening (Visit 1)must show no abnormalities suggestive of active TB infection as determined by a qualified medical specialist

   * Participants with a pre-existing demyelinating disorder such as multiple sclerosis or new onset seizures, unexplained sensory motor, or cognitive behavioral, neurological deficits, or significant abnormalities noted during screening
   * Participants with any unexplained symptoms suggestive of PML based on the targeted neurological assessment during the screening period
   * Participants with a transplanted organ. Skin grafts to treat pyoderma gangrenosum are allowed
   * Participants with a significant concurrent medical condition at the time of screening (Visit 1) or baseline (Visit 2), including, but not limited to, the following:

a. Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, GI [except disease under study], endocrine, cardiovascular, pulmonary, immunologic [eg, Felty's syndrome], or local active infection/infectious illness) that, in the investigator's judgment will substantially increase the risk to the subject if he or she participates in the study b. Cancer or history of cancer or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence) c. Presence of acute coronary syndrome (eg, acute myocardial infarction, unstable angina pectoris) within 24 weeks before screening (Visit 1) d. History of significant cerebrovascular disease within 24 weeks before screening (Visit 1)

* Participants who have had significant trauma or major surgery within 4 weeks before the screening (Visit 1), or with any major elective surgery scheduled to occur during the study.
* Participant with evidence of cirrhosis with or without decompensation (ie, esophageal varices, hepatic encephalopathy, portal hypertension, ascites)
* Participant with primary sclerosing cholangitis
* Participant with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) Note: if a subject tests negative for HBsAg, but positive for HBcAb, the subject would be considered eligible if no presence of hepatitis B virus (HBV) DNA is confirmed by HBV DNA polymerase chain reaction (PCR) reflex testing performed in the central laboratory
* Participant with chronic hepatitis C virus (HCV) (positive HCV antibody [HCVAb] and HCV RNA) Note: Participant who are HCVAb positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks prior to baseline])
* Participant with any of the following abnormalities in hematology and/or serum chemistry profiles during screening (Visit 1) Note: Screening laboratory tests, if the results are considered by the investigator to be transient and inconsistent with the subject's clinical condition, may be repeated once during the screening period for confirmation results must be reviewed for eligibility prior to the screening colonoscopy procedure

  1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels >=3.0 × the upper limit of normal (ULN)
  2. Total bilirubin level >=1.5 × ULN or >2.0 × ULN if the subject has a known documented history of Gilbert's syndrome
  3. Hemoglobin level less than or equal to(<=80) gram per liter(g/L) (8.0 g/deciliter[dL])
  4. Platelet count <=100× 10^9/L (100,000 cells/mm^3) or >=1000 × 10^9/L (1,000,000 cells/mm^3)*
  5. White blood cell count <=3.5 × 10^9/L (3500 cells/mm^3)
  6. Absolute neutrophil count <2 × 10^9/L (2000 cells/mm^3)
  7. Serum creatinine level >1.5 × ULN or estimated glomerular filtration rate <30 millilter per minute (mL/min)/173 meter square (m^2) based on the abbreviated Modification of Diet in RenalDisease Study Equation Note: if platelet count is <150,000 cells/mm3, a further evaluation should be performed to rule out cirrhosis, unless another etiology has already been identified
* Participant with known human immunodeficiency virus (HIV) infection based on documented history with positive serological test, or positive HIV serologic test at screening, tested at the site's local laboratory in accordance with country requirements or tested at the central laboratory Note: A documented negative HIV test within 6 months of screening is acceptable and does not need to be repeated
* With known human immunodeficiency virus (HIV) infection based on documented history with positive serological test, or positive HIV serologic test at screening, tested at the site's local laboratory in accordance with country requirements or tested at the central laboratory.
* Participants who have, or who have a history of (within 2 years before screening), serious psychiatric disease, alcohol dependency, or substance/drug abuse or dependency of any kind including abuse of medicinal marijuana (cannabis)

NOTE: The above Inclusion/Exclusion criteria are NOT exhaustive and other Inclusion/ Exclusion criteria as defined in the protocol may apply.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (145):
- United States (48):
  - Arizona Digestive Health Mesa - East, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - Clinedge - PPDS, Phoenix, Arizona
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Alliance Clinical Research-(Vestavia Hills), Poway, California
  - Care Access Research, San Pablo, San Pablo, California
  - Renaissance Research Medical Group, INC, Cape Coral, Florida
  - Gastro Florida, Clearwater, Florida
  - Alliance Medical Research LLC, Coral Springs, Florida
  - SIH Research, Kissimmee, Florida
  - Hi Tech and Global Research, LLc, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Pharma Research International Inc, Naples, Florida
  - Bayside Clinical Research - New Port Richey, New Port Richey, Florida
  - Accel Research Sites - St. Petersburg - ERN - PPDS, Pinellas Park, Florida
  - DBC Research, Tamarac, Florida
  - Infinite Clinical Trials, Atlanta, Georgia
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Loretto Hospital, Chicago, Illinois
  - IL Gastroenterology Group, Gurnee, Illinois
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - CroNOLA, LLC., Houma, Louisiana
  - DelRicht Clinical Research, LLC - ClinEdge - PPDS, New Orleans, Louisiana
  - Commonwealth Clinical Studies LLC, Brockton, Massachusetts
  - Winchester Gastroenterology Associates, Winchester, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - Mayo Clinic Health System - PPDS, Duluth, Minnesota
  - Minnesota Gastroenterology PA, Plymouth, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Encompass Care, North Las Vegas, Nevada
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Southtowns Gastroenterology, PLLC, Orchard Park, New York
  - Penn State Hershey Medical Group, State College, Pennsylvania
  - Digestive Health Associates of Texas, P.A.dba DHAT Research Institute, Garland, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - BI Research Center, Houston, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - Mid Atlantic Health Specialists, Galax, Virginia
- Argentina (2):
  - Fundación Favaloro, Buenos Aires
  - Hospital Privado Centro Médico de Córdoba, Córdoba
- Belgium (3):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - CHU Mouscron, Mouscron
- Clinical Center Banja Luka, Banja Luka, Bosnia and Herzegovina
- Bulgaria (9):
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment Eurohospital, Plovdiv
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Medical Center Convex EOOD, Sofia
  - Diagnostic Consultative Centre Mladost - M OOD, Varna
- Colombia (2):
  - Fundación Valle Del Lili, Cali, Valle del Cauca Department
  - IPS Centro Médico Julián Coronel S.A.S. - PPDS, Cali, Valle del Cauca Department
- Estonia (2):
  - OÜ LV Venter, Pärnu
  - West Tallinn Central Hospital, Tallinn
- Greece (5):
  - Ippokrateio General Hospital of Athens, Athens, Attica
  - University General Hospital of Heraklion, Heraklion
  - Iatriko Palaiou Falirou, Paliao Faliro
  - University General Hospital of Patras, Pátrai
  - Euromedica - PPDS, Thessaloniki
- Hungary (8):
  - Bekes Megyei Kozponti Korhaz, Békéscsaba
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - ENDOMEDIX Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Mohacsi Korhaz, Mohács
  - Tolna Megyei Balassa János Kórház, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- St Vincent's University Hospital, Dublin, Ireland
- Japan (11):
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Medical Corporation Aoyama Clinic, Kobe, Hyôgo
  - Hyogo College of Medicine, Nishinomiya-shi, Hyôgo
  - Kunimoto Hospital, Asahikawa
  - Chiinkai Dojima General & Gastroenterology Clinic, Osaka
  - Kinshukai Infusion Clinic, Osaka
  - Yodogawa Christian Hospital, Osaka
  - Toho University Sakura Medical Center, Sakura
  - Dokkyo Medical University Hospital, Shimotsuga-gun
  - Nihonbashi Egawa Clinic, Tokyo
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Ôita
- Lebanon (2):
  - Al Zahraa University Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Mexico (8):
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Health Pharma Professional Research S.A de C.V., Mexico City, Mexico City
  - Clinica de Higado y Gastroenterologia Integral, S.C., Cuernavaca, Morelos
  - JM Research S.C, Cuernavaca, Morelos
  - Accelerium, S. de R.L. de C.V., Monterrey, Nuevo León
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Centro de Investigacion Clinica Acelerada, S.C., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
- New Zealand (3):
  - Dunedin Hospital, Dunedin, South Island
  - Wellington Hospital, Newtown, Wellington Region
  - Waikato Hospital, Hamilton
- Portugal (3):
  - Hospital da Luz, Lisbon, Lisbon District
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Centro Hospitalar do Algarve - Hospital de Portimao, Portimão
- Slovakia (2):
  - KM Management, spol. s r.o., Nitra
  - Gastro LM, s.r.o., Prešov
- South Korea (11):
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeonggido
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (9):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid, Madrid, Communidad Delaware
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Centro Medico Teknon - Grupo Quironsalud, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Mersin University Medical Faculty, Mersin
- Ukraine (13):
  - Regional Municipal Non-profit Enterprise "Chernivtsi Regional Clinical Hospital", Chernivtsi, Chernivtsi Oblast
  - Municipal Nonprofit Enterprise CCH #2 n.a. prof. O.O. Shalimov of Kharkiv City Council, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv, Kyïv
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - Municipal Nonprofit Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Municipal Non-profit Enterprise Kherson City Clinical Hospital named after Ye.Ye. Karabelesh, Kherson
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv
  - Medical Center OK!Clinic+LLC International Institute of Clinical Research, Kyiv
  - Medical Center of LLC Medical Center Dopomoga-Plus, Kyiv
  - Communal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Hospital, Kyiv
  - Municipal Nonprofit Enterprise Lviv Clinical Emergency Care Hospital, Lviv
  - Communal Non-Commercial Enterprise "Vinnytsia City Clinical Hospital No1", Vinnytsia
  - MNPE City Hospital No. 6 of Zaporizhzhia City Council, Zaporizhzhia

REFERENCES:
- [Derived] Vermeire S, Danese S, Sandborn WJ, Schreiber S, Hanauer S, D'Haens G, Nagy P, Thakur M, Bliss C, Cataldi F, Goetsch M, Gorelick KJ, Reinisch W. Efficacy and Safety of the Anti-mucosal Addressin Cell Adhesion Molecule-1 Antibody Ontamalimab in Patients with Moderate-to-Severe Ulcerative Colitis or Crohn's Disease. J Crohns Colitis. 2024 May 31;18(5):708-719. doi: 10.1093/ecco-jcc/jjad199. PMID 38096402
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe54db2bf003ab47918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 sites in the Unites States, Belgium, Bosnia and Herzegovina, Colombia, Hungary, Japan, Mexico, Slovakia, Republic of Korea, Spain and Ukraine between 17 July 2018 (first participant first visit) and 18 August 2020 (last participant last visit).
Pre-assignment Details: A total of 34 participants were enrolled into the study, of which 27 participants completed the study. Other secondary outcome measures were not analyzed due to early discontinuation of the study for reasons unrelated to safety.
Groups:
- Placebo: Participants received ontamalimab matching-placebo, injection, subcutaneously using a prefilled syringe on Week 0 (Day 1), Week 4, Week 8, and Week 12 in a 16-week treatment period.
- Ontamalimab 25 mg: Participants received ontamalimab 25 milligram (mg), injection, subcutaneously using a prefilled syringe on Week 0 (Day 1), Week 4, Week 8, and Week 12 in a 16-week treatment period.
- Ontamalimab 75 mg: Participants received ontamalimab 75 mg, injection, subcutaneously using a prefilled syringe on Week 0 (Day 1), Week 4, Week 8, and Week 12 in a 16-week treatment period.
Period: Overall Study
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Started | 6 | 15 | 13
Completed | 4 | 12 | 11
Not Completed | 2 | 3 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who had received at least 1 dose of investigational product (IP).
Groups:
- Ontamalimab 25 mg: Participants received ontamalimab 25 mg, injection, subcutaneously using a prefilled syringe on Week 0 (Day 1), Week 4, Week 8, and Week 12 in a 16-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg | Total
Number analyzed (Participants) | 6 | 15 | 13 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.60) | 37.5 (10.20) | 39.1 (12.74) | 39.0 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 5 | 15
  Male | 4 | 7 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 4 | 14 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 1 | 2
  White | 3 | 12 | 11 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Remission Based on 2-item Patient-reported Outcome (PRO) at Week 16
Description: Clinical remission was defined by 2-item PRO subs-cores of average worst daily abdominal pain less than or equal to (<=) 3 (based on 11 point numerical rating scale [NRS] ranging from 0 [no pain] to 10 [worst imaginable pain]); and average daily stool frequency <=2 of type 6/7 (very soft stools/liquid stools) as per the Bristol Stool Form Scale (BSFS) over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like a sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, a mushy stool), 7 (watery, no solid pieces, entirely liquid). Participants with missing data at Week 16 or discontinuation before Week 16 were considered failures. Number of participants with clinical remission were reported.
Time Frame: At Week 16
Population: The full analysis set (FAS) consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 3 | 5 | 5

2. Primary Outcome: Number of Participants With Endoscopic Response at Week 16
Description: Endoscopic response was defined as a decrease in Simple Endoscopic Score for Crohn's disease (SES-CD) of at least 25 percent (%) from baseline. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Participants with missing data at Week 16 or who discontinued before Week 16 were considered failures. Number of participants with endoscopic response were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 2 | 10 | 10

3. Secondary Outcome: Number of Participants With Clinical Remission Based on Crohn's Disease Activity Index (CDAI) Score at Week 16
Description: Clinical remission was defined as a CDAI score of <150. CDAI assesses CD based on clinical signs/symptoms such as number of liquid stools, intensity of abdominal pain, general well-being (subjective), and presence of complications, use of antidiarrheal, presence of abdominal mass, physical examination and hematocrit (objective). CDAI score is equal to sum of weighted scores for subjective and objective items which range from 0-149 points: asymptomatic remission, 150-220 points: mild to moderate active CD, 221-450 points: moderate to severe active CD, >451 points: severely active to fulminant disease. Higher score indicating more severity. Number of participants with clinical remission as measured by CDAI were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 4 | 8 | 6

4. Secondary Outcome: Number of Participants With Enhanced Endoscopic Response at Week 16
Description: Enhanced endoscopic response was defined as a decrease in SES-CD by matching segments of at least 50% from baseline. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Participants with missing data at Week 16 or who discontinued before Week 16 were considered non-responders. Number of participants with enhanced endoscopic response were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 2 | 5 | 3

5. Secondary Outcome: Number of Participants With Clinical Remission Based on 2-item PRO With 4-point Scale for Abdominal Pain at Week 16
Description: Clinical remission was defined by 2-item PRO subs-cores of average daily abdominal pain <=1 (based on the 4 point scale, with scores ranging from 0 [none] to 3 [severe]) over the 7 most recent days and average daily stool frequency <=3 of type 6/7 (very soft stools/liquid stools) as per the BSFS over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like a sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, a mushy stool), 7 (watery, no solid pieces, entirely liquid). Participants with missing data at Week 16 or who discontinued before Week 16 were considered failures. Number of participants with enhanced endoscopic response were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 3 | 6 | 6

6. Secondary Outcome: Number of Participants With Clinical Response Based on 2-item PRO With 2 Criteria at Week 16
Description: Clinical response was measured by 2-item PRO and defined as meeting at least 1 of the following 2 criteria: 1)A decrease of greater than or equal to (>=) 30% and at least 2 points from baseline in the average daily worst abdominal pain over the 7 most recent days, with the average daily stool frequency of type 6/7 (very soft stools/liquid stools) either a) not worsening from baseline and/or b) average daily stool frequency <=2 of type 6/7 as per the BSFS over the 7 most recent days; 2)A decrease of >=30% from baseline in the average daily stool frequency of type 6/7 (very soft stools/liquid stools) as per the BSFS over the 7 most recent days, with the average daily worst abdominal pain either a) not worsening from baseline and/or b) worst daily abdominal pain <=3 (based on 11-point NRS) over the 7 most recent days. Participants with missing data at Week16 or who discontinued before Week 16 were considered failures. Number of participants with clinical response were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 5 | 11 | 8

7. Secondary Outcome: Number of Participants With Clinical Remission Based on 2-Item PRO With Endoscopic Response at Week 16
Description: Clinical remission was defined by 2-item PRO subs-cores of average worst daily abdominal pain <=3 (based on 11 point NRS ranging from 0 [no pain] to 10 [worst imaginable pain]) over the 7 most recent days and average daily stool frequency <=2 of type 6/7 (very soft stools/liquid stools) as per BSFS ranging from type 1 (separate hard lumps-like stools) to type 7 (entirely liquid stools) over the 7 most recent days. Endoscopic response was defined as a decrease in SES CD of at least 25% from baseline. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Participants with missing data at Week 16 or who discontinued before Week 16 were considered failures. Number of participants with clinical remission and endoscopic response were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 1 | 4 | 5

8. Secondary Outcome: Number of Participants With Complete Endoscopic Healing at Week 16
Description: Clinical remission was defined by 2-item PRO subs-cores of average worst daily abdominal pain <=3 (based on 11 point NRS ranging from 0 [no pain] to 10 [worst imaginable pain]) over the 7 most recent days and average daily stool frequency <=2 of type 6/7 (very soft stools/liquid stools) as per BSFS ranging from type 1 (separate hard lumps-like stools) to type 7 (entirely liquid stools) over the 7 most recent days. Endoscopic response was defined as a decrease in SES CD of at least 25% from baseline. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease. Participants with missing data at Week 16 or who discontinued before Week 16 were considered failures. Number of participants with complete endoscopic healing were reported.
Time Frame: At Week 16
Population: The FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 15 | 13
Participants | 1 | 3 | 2

9. Secondary Outcome: Number of Participants With Clinical Response as Measured by CDAI-100 at Week 16
Description: Clinical response was measured by at least a 100-point reduction in the CDAI from baseline (CDAI-100 response). CDAI assesses CD based on clinical signs/symptoms such as number of liquid stools, intensity of abdominal pain, general well-being (subjective), and presence of complications, use of antidiarrheal, presence of abdominal mass, physical examination and hematocrit (objective). CDAI score is equal to sum of weighted scores for subjective and objective items which range from 0-149 points: asymptomatic remission, 150-220 points: mild to moderate active CD, 221-450 points: moderate to severe active CD, >451 points: severely active to fulminant disease. Higher score indicating more severity.
Time Frame: At Week 16
Population: Study terminated early for reasons unrelated to safety. Hence, for this outcome measure, the planned data collection and analysis was not performed.
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinical Response as Measured by CDAI-70 at Week 16
Description: Clinical response was measured by at least a 70-point reduction in the CDAI from baseline (CDAI-70 response). CDAI assesses CD based on clinical signs/symptoms such as number of liquid stools, intensity of abdominal pain, general well-being (subjective), and presence of complications, use of antidiarrheal, presence of abdominal mass, physical examination and hematocrit (objective). CDAI score is equal to sum of weighted scores for subjective and objective items which range from 0-149 points: asymptomatic remission, 150-220 points: mild to moderate active CD, 221-450 points: moderate to severe active CD, >451 points: severely active to fulminant disease. Higher score indicating more severity.
Time Frame: At Week 16
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinical Remission Over Time
Description: Clinical remission was defined by 2-item PRO subs-cores of average worst daily abdominal pain (based on 11 point NRS ranging from 0 [no pain] to 10 [worst imaginable pain]); and average daily stool frequency of type 6/7 (very soft stools/liquid stools) as per BSFS over the 7 most recent days. BSFS ranges from 1 (separate hard lumps, hard to pass), 2 (sausage-shaped, but lumpy), 3 (like a sausage but with cracks on the surface), 4 (like a sausage or snake, smooth and soft), 5 (soft blobs with clear-cut edges), 6 (fluffy pieces with ragged edges, a mushy stool), 7 (watery, no solid pieces, entirely liquid).
Time Frame: At Week 16
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Individual and Total Sign/Symptom Score Based on Participant Daily Electronic Diary (E-diary) Entries
Description: CD clinical signs and symptoms includes total stool frequency, rectal bleeding frequency, rectal urgency frequency, nausea severity, vomiting frequency, and rectal incontinence frequency.
Time Frame: Baseline and at Week 16
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Endoscopic Healing at Week 16
Description: Endoscopic healing was measured by SES-CD <=4 and at least 2-point reduction versus baseline and no sub-score >1 in any individual variable. The SES-CD considers ileum, right colon, transverse colon, left colon, rectum in terms of: size of ulcers, ulcerated surface, affected surface and presence of narrowing. Each graded from 0-3. Scale ranges from 0-56 with a higher score indicating greater severity of disease.
Time Frame: At Week 16
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total (Absolute) Score at Weeks 8, 12 and 16
Description: The IBDQ is a psychometrically validated PRO instrument for measuring the disease-specific health-related quality of life (HRQL) in participants with IBD, including CD. The IBDQ consists of 32 items, which are grouped into 4 domains and scored as: bowel function (10 to 70), systemic symptoms (5 to 35), emotional status (12 to 84), and social function (5 to 35). The total IBDQ score ranges from 32 to 224. For the total score and each domain, a higher score indicates better HRQL. A score of at least 170 corresponds to clinical remission and an increase of at least 16 points is considered to indicate a clinically meaningful improvement.
Time Frame: Baseline, Weeks 8, 12 and 16
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36) Scores at Week 16
Description: The SF-36, version 2 is a generic quality-of-life instrument that has been widely used to assess HRQL of participants. The SF-36 consists of 36 items that are aggregated into 8 multi-item scales (physical functioning, role - physical, bodily pain, general health, vitality, social functioning, role - emotional, and mental health), with scores ranging from 0 to 100. Higher scores indicate better HRQL.
Time Frame: Baseline, Week 16
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Based on Incidence of All-cause Hospitalizations
Description: Incidence of all cause hospitalizations was planned to be assessed.
Time Frame: Baseline up to Week 32
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Number of Participants Based on Total Inpatient Days
Description: Total inpatient days were planned to be assessed.
Time Frame: Baseline up to Week 32
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Based on Incidence of CD-related Surgeries and Other Surgical Procedures
Description: Incidence of CD-related surgeries and other surgical procedures were planned to be recorded.
Time Frame: Baseline up to Week 32
Population: as for outcome 9
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening up to safety follow-up period (Week 32)
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/15 | 2/13
Other Adverse Events (participants affected / at risk) | 6/6 | 6/15 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Ontamalimab 25 mg (N=15) | Ontamalimab 75 mg (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Ontamalimab 25 mg (N=15) | Ontamalimab 75 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pain threshold decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated as the sponsor discontinued the ontamalimab clinical trial program in ulcerative colitis and CD for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03566823/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03566823/SAP_001.pdf